CLINICAL TRIAL: NCT00633763
Title: PET-CT Scan Method to Monitor Pancreatic B-Cell Loss in Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: K. George Chandy, Professor, Department of Physiology and Biophysics, UC Irvine
Other Study IDs: 2007-5785
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Diagnostic; PET/CT imaging of pancreas; Detecting pancreatic beta cell loss during diabetes
MeSH Terms: conditions — Disease | interventions — N-((1-allyl-2-pyrrolidinyl)methyl)-5-(3-fluoropropyl)-2,3-dimethoxybenzamide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Healthy individuals with normal C-peptide levels following i.v. glucagon challenge. These individuals will be administered 18F-fallypride and then subjected to PET-CT scanning of the pancreas and brain. The subject will be positioned in the PET/CT scanner and a low-dose CT (15-20 secs) of the abdomen carried out (with subjects breathing normally). A 30-min PET acquisition will then be started (three 10 min static frames or one 30 min static frame). The subject will then be repositioned for a low-dose CT scan of the head (15-20 secs) following which a 20-min PET acquisition will then be started (two 10 min static frames or one 20 min static frame).
  Interventions: Drug: 18F-fallypride
- 2: Patients with longstanding T1DM and <20% C-peptide levels following i.v. glucagon challenge will be consented. 18F-Fallypride injected intravenously and subjects allowed to wait for approx 1 hr for the uptake.(b) Subject positioned in the PET/CT scanner and a low-dose CT (15-20 secs) of the abdomen (pancreas) carried out (with subjects breathing normally).(c) A 30-min PET acquisition will then be started (three 10 min static frames or one 30 min static frame).(d) Subject repositioned for a low-dose CT scan of the head (15-20 secs).(e) A 20-min PET acquisition will then be started (two 10 min static frames or one 20 min static frame).(f) End of PET/CT scanning procedures. Subject taken out of the scanner.
  Interventions: Drug: 18F-fallypride

INTERVENTIONS:
Drug: 18F-fallypride — Single bolus i.v. injection 60 minutes before PET-CT scanning. Maximum activity per single administration 5 mCi; maximum amount of drug per administration <10 micrograms.
Drug: 18F-fallypride — I.v. bolus maximum activity per single administration 5 mCi; maximum amount of drug per administration <10 micrograms.

SUMMARY:
The pancreas is an organ that plays major roles in the digestion of food. A part of the pancreas called islet beta-cells produces insulin, which regulates the amount of glucose (a sugar) present in the blood at all times. Type-1 Diabetes Mellitus (T1DM), an autoimmune disorder characterized by destruction of pancreatic islet beta-cells (the cells that produce insulin), affects at least a million individuals in the US alone. In T1DM, a type of white blood cells called T lymphocytes attacks and destroys the pancreatic islet beta-cells, leading to a loss of insulin, an increase in blood glucose, and a dependence on insulin injections for survival. Despite rigorous control of blood sugar, the majority of diabetic patients develop serious complications including retinopathy, nephropathy, neuropathy, microangiopathy and strokes.

Non-invasive methods to monitor pancreatic beta-cell loss associated with type-1 diabetes mellitus (T1DM) could improve early diagnosis, provide tools to measure responsiveness to new therapies, and evaluate the efficiency of pancreatic transplantation and graft survival.

Our goal is to develop a non-invasive PET-CT imaging method based on binding of a molecule (18F-fallypride) for tracking beta-cell loss during the progression of T1DM. In preliminary studies we demonstrated specific binding of 18F-fallypride to D2 receptors in rat pancreatic sections and we demonstrated that the loss of pancreatic beta cells in streptozotocin-treated rats was associated with a corresponding decrease in 18F-fallypride binding to pancreatic sections. A preliminary 18F-fallypride PET-CT study done by a collaborator in Ohio on a healthy volunteer, revealed 18F-fallypride-uptake by the pancreas that was distinguishable from surrounding tissues. Aim-1 of our project will measure the variability of 18F-fallypride PET-scanning of the pancreas in six healthy volunteers scanned twice with an interval of 4-6 weeks. In Aim-2 of our project, we will compare fallypride PET-CT scans of 12 patients with long-standing T1DM (nearly all beta cells destroyed) with 12 age- and sex-matched healthy volunteers. If we are able to distinguish between the two groups, we will in future (a) optimize the method so as to be able to detect a 20-30% loss of beta cells, and (b) perform PET-CT studies in new-onset T1DM patients and in at-risk first degree relatives of T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* T1DM patients that are over 18 years of age, have had T1DM for greater than 5 years and show a greater than 80% reduction in C-peptide blood levels following intravenous glucagon injection are eligible to participate in this study.
* Healthy controls that are over 18 years of age, show normal C-peptide blood levels following intravenous glucagon injection, and are age- and sex-matched with one of the T1DM patients included in the study, are eligible to participate in this study.

Exclusion Criteria:

* T1DM patients or healthy controls that are not over 18 years of age are not eligible to participate in this study.
* Pregnant females are not eligible to participate in this study because there is a chance PET/CT scans might be risky for the developing baby. Females physically capable of getting pregnant will be required to get a urine pregnancy test at no cost before each of the PET/CT scans. If the pregnancy test is positive, the T1DM patient or healthy control will be excluded from the study. The consent form describes the risks in detail and the need for women of childbearing age to undergo a pregnancy test.
* Subjects with a history of psychiatric illness, substance abuse history, clinically significant head trauma, active neurological disease, cardiovascular disease, liver disease or renal impairment, claustrophobia ((very upset and afraid of being in a small space) are not eligible for the study. Dr. Ping Wang will use the subjects history, blood chemistry, to identify individuals with cardiovascular disease, liver disease, or renal impairment.
* T1DM patients with C-peptide levels following intravenous glucagon injection that are not reduced greater than 80% are not eligible for the study.
* Healthy volunteers with C-peptide levels following intravenous glucagon injection that are reduced greater than 20% compared to established control values are not eligible for the study.
* To determine if it is safe to do the procedure, T1DM patients and healthy volunteers will be expected to tell the researchers about any radiation exposure the individual may have had (including diagnostic or treatment x-rays), and any history of head injury, kidney or bladder disease, or any other serious medical conditions.
* T1DM patients and healthy volunteers will be expected to tell the researchers if they have surgical clips or metallic prostheses (i.e., replacement body parts, such as a hip joint) or a pacemaker or other pieces of metal in the body (shrapnel, metal filings, etc.).
* Patients with history of alcoholism or significant alcohol consumption will be excluded from the study.
* The consent form will be English, and non-English speakers will therefore be excluded from the study.
* Pregnant women are excluded because 18F-fallypride is a radioactive substance , which will be injected into the patient and could be hazardous to the fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Joslin Diabetes Clinic at the University of California Irvine, age-matched controls will be obtained from Orange County California.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Difference in fallypride binding in the pancreas of long-standing T1DM patients versus healthy controls | At the end of the study when 12 controls and 12 patients have been studied.

CONTACTS AND LOCATIONS:
Overall Officials: George K Chandy, MD, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States